CLINICAL TRIAL: NCT06525974
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Febuxostat in Patients With Ulcerative Colitis Treated With Mesalamine
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohammed El-kabbary Hasan Diab, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.24.04.2758
Record Dates: First submitted 2024-06-29; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Febuxostat; Mesalamine
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Febuxostat; Mesalamine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Mesalamine group) (Active Comparator): Control group (Mesalamine group, n =23) who will receive 1 g mesalamine three times daily for 3 months.
  Interventions: Drug: Mesalamine
- Experimental group (Febuxostat group) (Experimental): Experimental group (Febuxostat group, n = 23) which will receive the standard treatment for UC plus 40 mg febuxostat once daily for 3 months.
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — 40mg of Febuxostat once daily
  Arms: Experimental group (Febuxostat group)
Drug: Mesalamine — 1 g mesalamine three times daily for 3 months.
  Arms: Control group (Mesalamine group)

SUMMARY:
Evaluation the possible efficacy and safety of febuxostat in patients with ulcerative colitis treated with mesalamine.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a sub-category of inflammatory bowel diseases (IBD) that causes mucosal inflammation in the rectum and lower colon. Although the exact pathogenesis of ulcerative colitis remains unclear, potential risk factors include altered immune responses, overactive immune response toward commensal microflora, genetic susceptibility, and environmental factors that have been considered as potential risk factors for UC .

The pathogenesis of UC consists of immuno-inflammatory pathways related to the multiple components of the intestine, including the epithelial barrier, dysregulation of immunological responses, leukocyte recruitment, and genetic factors. The understanding of immuno-inflammatory pathways of UC might lead to the development of a specific therapy and/or a novel treatment that could be more efficient .

Mesalazine (also known as mesalamine or 5- amino salicylic acid, 5-ASA) has a well-established role in UC management. It is the first line therapy for mild to moderate UC and it is considered the cornerstone in the management of UC. The mechanism of action of mesalazine is diverse. It acts locally on colonic mucosa and reduces inflammation by several anti-inflammatory processes .

Febuxostat (FXT) is a medication used in management hyperuricemia espicially in gout, a condition characterized by joints pain as result of deposition of uric acid crystals due to elevated urate blood levels. It's a non-purine selective xanthine oxidase inhibitor. Xanthin oxidase is an enzyme that plays a main role in production of uric acid from xanthine and hypoxanthine.

Furthermore, there is no need for dose modification of FXT in case of renal impairment and so it's great choice for many patients as it may exhibit renal protective effect and delay progression of kidney injury and according to Zhou H et al. FXT appears to be well tolerated in healthy population who has normal serum uric acid levels with no serious adverse events were reported .

Lately, febuxostat's spectrum of use has expanded over hyperuricemia management as result of it's ability of amelioration oxidative stress and regulation inflammatory response due to pro -inflammatory cytokines modulation.

Keyvan Amirshahrokhi and El-Mahdy NA et al. inspected the potential of FXT in mitigating ulcerative colitis in mice. The findings from those studies suggest that febuxostat may exert anti- inflammatory effects in the context of ulcerative colitis. Febuxostat's anti- inflammatory effects in ulcerative colitis may be linked to its inhibition of the nuclear factor kappa B (NF-κB) signaling pathway, a key regulator of inflammation. This inhibition can reduce the production of proinflammatory cytokines, contributing to its anti-inflammatory properties .

Although, preclinical studies in animal models are promising, translating these results into clinical applications is necessary to evaluate the safety and efficacy of FXT in managing UC in human.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Both male and female will be included.
* Mild and moderate UC patients diagnosed and confirmed by endoscope.
* Patient treated with 5-aminosalislic acid (mesalamine).

Exclusion Criteria:

* Patients with severe UC.
* Significant liver and kidney function abnormalities.
* Diabetic patients.
* Patients with Colorectal cancer patients.
* Patients taking rectal or systemic steroids.
* Patients on immunosuppressants or biological therapies.
* Addiction to alcohol and / or drugs.
* Known allergy to the studied medications.
* History of complete or partial colectomy.
* Patients with congestive heart failure, other heart disease (Arrhythmia, ischemic heart disease including angina and myocardial infarction).
* Patients with other inflammatory diseases and active infection.
* Patients with stressful condition (COPD, morbid obesity).
* Patients with liver disease.
* Patients with thrombocytopenia and neutropenia.
* Pregnant or lactating females.
* Patients were treated with mercaptopurine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of disease activity using Partial Mayo Scoring Index (PMSI) assessment for Ulcerative Colitis Activity. | 3 months
  It depends on three items: stool frequency, rectal bleeding (blood in stool) and Physician's Global Assessment. Each item has a score from 0 to 3 and total PMSI is the sum of scores for the three items.
Health-related quality of life (HRQOL) using the short inflammatory bowel disease questionnaire . | 3 months
  Short Inﬂammatory Bowel Disease Ques-tionnaire (SIBDQ) version became widely known and is currently used worldwide both in clinical practice and clinical research. SIBDQ comprises a total of 10 questions grouped into four diﬀerent dimensions: social, bowel, emotional, and systemic [6, 7]. Each question is scored by a 7-point Likert scale, ranging from 1 (a severe problem) to 7 (not a problem at all), giving an absolute SIBDQ score ranging from 10 (poor HRQoL) to 70 (opti-mal HRQoL). A SIBDQ score below 50 was considered as poor QoL.there are no validated cut-oﬀs for the dif-ferent dimensions' scores. Hence, higher scores indicate a better HRQoL concerning that speciﬁc domain.Although patient-reported outcomes are highly valu-able for better patient care, patient responses to HRQoL instruments can be impacted by underlying cultural trends

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Abdel-Wahab BA, El-Shoura EAM, Shafiuddin Habeeb M, Zafaar D. Febuxostat alleviates Arsenic Trioxide-Induced renal injury in Rats: Insights on the crosstalk between NLRP3/TLR4, Sirt-1/NF-kappaB/TGF-beta signaling Pathways, and miR-23b-3p, miR-181a-5b expression. Biochem Pharmacol. 2023 Oct;216:115794. doi: 10.1016/j.bcp.2023.115794. Epub 2023 Sep 7. PMID 37689273
- [Background] Amirshahrokhi K. Febuxostat attenuates ulcerative colitis by the inhibition of NF-kappaB, proinflammatory cytokines, and oxidative stress in mice. Int Immunopharmacol. 2019 Nov;76:105884. doi: 10.1016/j.intimp.2019.105884. Epub 2019 Sep 6. PMID 31499267
- [Background] Cicero AFG, Fogacci F, Kuwabara M, Borghi C. Therapeutic Strategies for the Treatment of Chronic Hyperuricemia: An Evidence-Based Update. Medicina (Kaunas). 2021 Jan 10;57(1):58. doi: 10.3390/medicina57010058. PMID 33435164
- [Background] El-Mahdy NA, Saleh DA, Amer MS, Abu-Risha SE. Role of allopurinol and febuxostat in the amelioration of dextran-induced colitis in rats. Eur J Pharm Sci. 2020 Jan 1;141:105116. doi: 10.1016/j.ejps.2019.105116. Epub 2019 Oct 23. PMID 31654756
- [Background] Elsisi AEE, Sokar SS, Shalaby MF, Abu-Risha SE. Nephroprotective effects of febuxostat and/or mirtazapine against gentamicin-induced nephrotoxicity through modulation of ERK 1/2, NF-kappaB and MCP1. Expert Rev Clin Pharmacol. 2021 Aug;14(8):1039-1050. doi: 10.1080/17512433.2021.1933435. Epub 2021 Jun 9. PMID 34030558
- [Background] Fukui T, Maruyama M, Yamauchi K, Yoshitaka S, Yasuda T, Abe Y. Effects of Febuxostat on Oxidative Stress. Clin Ther. 2015 Jul 1;37(7):1396-401. doi: 10.1016/j.clinthera.2015.03.026. Epub 2015 Apr 23. PMID 25913922
- [Background] Hao G, Duan W, Sun J, Liu J, Peng B. Effects of febuxostat on serum cytokines IL-1, IL-4, IL-6, IL-8, TNF-alpha and COX-2. Exp Ther Med. 2019 Jan;17(1):812-816. doi: 10.3892/etm.2018.6972. Epub 2018 Nov 15. PMID 30651867
- [Background] Irvine EJ, Zhou Q, Thompson AK. The Short Inflammatory Bowel Disease Questionnaire: a quality of life instrument for community physicians managing inflammatory bowel disease. CCRPT Investigators. Canadian Crohn's Relapse Prevention Trial. Am J Gastroenterol. 1996 Aug;91(8):1571-8. PMID 8759664
- [Background] Kanji T, Gandhi M, Clase CM, Yang R. Urate lowering therapy to improve renal outcomes in patients with chronic kidney disease: systematic review and meta-analysis. BMC Nephrol. 2015 Apr 19;16:58. doi: 10.1186/s12882-015-0047-z. PMID 25928556
- [Background] Kim YE, Ahn SM, Oh JS, Kim YG, Lee CK, Yoo B, Hong S. Febuxostat dose requirement according to renal function in patients who achieve target serum urate levels: A retrospective cohort study. Joint Bone Spine. 2024 Mar;91(2):105668. doi: 10.1016/j.jbspin.2023.105668. Epub 2023 Nov 29. PMID 38036062
- [Background] Kobayashi T, Siegmund B, Le Berre C, Wei SC, Ferrante M, Shen B, Bernstein CN, Danese S, Peyrin-Biroulet L, Hibi T. Ulcerative colitis. Nat Rev Dis Primers. 2020 Sep 10;6(1):74. doi: 10.1038/s41572-020-0205-x. PMID 32913180
- [Background] Sarhan II, Abdellatif YA, Saad RE, Teama NM. Renoprotective effect of febuxostat on contrast-induced acute kidney injury in chronic kidney disease patients stage 3: randomized controlled trial. BMC Nephrol. 2023 Mar 22;24(1):65. doi: 10.1186/s12882-023-03114-4. PMID 36949408
- [Background] Sloka J, Madej M, Strzalka-Mrozik B. Molecular Mechanisms of the Antitumor Effects of Mesalazine and Its Preventive Potential in Colorectal Cancer. Molecules. 2023 Jun 29;28(13):5081. doi: 10.3390/molecules28135081. PMID 37446747
- [Background] Solitano V, D'Amico F, Fiorino G, Paridaens K, Peyrin-Biroulet L, Danese S. Key Strategies to Optimize Outcomes in Mild-to-Moderate Ulcerative Colitis. J Clin Med. 2020 Sep 8;9(9):2905. doi: 10.3390/jcm9092905. PMID 32911840
- [Background] Sturm A, Maaser C, Calabrese E, Annese V, Fiorino G, Kucharzik T, Vavricka SR, Verstockt B, van Rheenen P, Tolan D, Taylor SA, Rimola J, Rieder F, Limdi JK, Laghi A, Krustins E, Kotze PG, Kopylov U, Katsanos K, Halligan S, Gordon H, Gonzalez Lama Y, Ellul P, Eliakim R, Castiglione F, Burisch J, Borralho Nunes P, Bettenworth D, Baumgart DC, Stoker J; European Crohn's and Colitis Organisation [ECCO] and the European Society of Gastrointestinal and Abdominal Radiology [ESGAR]. ECCO-ESGAR Guideline for Diagnostic Assessment in IBD Part 2: IBD scores and general principles and technical aspects. J Crohns Colitis. 2019 Mar 26;13(3):273-284. doi: 10.1093/ecco-jcc/jjy114. No abstract available. PMID 30137278
- [Background] Tatiya-Aphiradee N, Chatuphonprasert W, Jarukamjorn K. Immune response and inflammatory pathway of ulcerative colitis. J Basic Clin Physiol Pharmacol. 2018 Dec 19;30(1):1-10. doi: 10.1515/jbcpp-2018-0036. PMID 30063466
- [Background] Zhou H, Zheng Y, Wu G, Hu X, Zhai Y, Iv D, Liu J, Wu L, Shentu J. Pharmacokinetics and tolerability of febuxostat after oral administration in healthy Chinese volunteers: a randomized, open-label, singleand multiple-dose three-way crossover study. Int J Clin Pharmacol Ther. 2016 Feb;54(2):115-24. doi: 10.5414/CP202394. PMID 26636422